CLINICAL TRIAL: NCT03426345
Title: A 12-week, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of Relamorelin in Patients With Diabetic Gastroparesis
Brief Title: Study to Evaluate the Safety and Efficacy of Relamorelin in Participants With Diabetic Gastroparesis Study 02
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Relamorelin program is being terminated solely based on a business decision
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLM-MD-02; 2017-002177-20 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Following a 2-week placebo run-in, participants received placebo-matching relamorelin injected subcutaneously twice daily for up to 12 weeks.
  Interventions: Drug: Placebo
- Relamorelin 10 μg (Experimental): Following a 2-week placebo run-in, participants received relamorelin 10 micrograms (μg) injected subcutaneously twice daily for up to 12 weeks.
  Interventions: Drug: Relamorelin

INTERVENTIONS:
Drug: Placebo — Placebo injected subcutaneously twice daily.
  Arms: Placebo
Drug: Relamorelin — Relamorelin 10 μg injected twice daily for 12 weeks.
  Arms: Relamorelin 10 μg

SUMMARY:
This study will evaluate the safety and efficacy of relamorelin compared to placebo in participants with diabetic gastroparesis. Participants will report daily severity scores of their diabetic gastroparesis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 or Type 2 diabetes mellitus
* Meet the per protocol criteria of diabetic gastroparesis
* Compliance with diary
* Compliance with the per protocol study treatment dosing instructions

Exclusion Criteria:

* Currently receiving nutrition intravenously, by nasogastric tube, or other feeding tube
* Actively experiencing anorexia nervosa, binge-eating, bulimia or other eating disorder at the time of Screening (Visit 1)
* Diagnosis of Celiac Disease, also a history of non-celiac gluten sensitivity
* History of gastrointestinal disorders that may be similar to gastroparesis
* Functional dyspepsia diagnosed before the diagnosis of diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw (Wes) Bochenek, MD, PhD, Study Director — Allergan
Locations (240):
- United States (114):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Synexus Clinical Research US - Simon Williamson Clinic, Birmingham, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Synexus Clinical Research US, Inc., Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Unity Health - Searcy Medical Center, Searcy, Arkansas
  - GW Research Inc., Chula Vista, California
  - Diagnamics Inc., Encinitas, California
  - Fresno Clinical Research Center, Fresno, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Angel City Research Inc., Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - Stanford Hospital, Digestive Health Clinic, Palo Alto, California
  - TriWest Research Associates, Poway, California
  - Optimal Research California, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - New Hope Research Development, Whittier, California
  - Synexus Clinical Research US, Inc. - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Gastroenterology Associates of Fairfield County, P.C., Bridgeport, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - ALL Medical Research LLC, Cooper City, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - Vida Clinical Trials, Homestead, Florida
  - Sanchez Clinical Research, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Synexus, Pinellas Park, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gwinnett Research Institute, LLC, Buford, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Clinical Research Consultants of Atlanta, Suwanee, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - American Research, LLC, Jeffersonville, Indiana
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - Health Science Research Center, Pratt, Kansas
  - WestGlen Gastrointestinal Consultants, Shawnee Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Via Christi Clinic, PA, Wichita, Kansas
  - Tri-State Gastroenterology, Crestview Hills, Kentucky
  - WK Physicians Network, Bossier City, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Clinical Trials of America, Inc., West Monroe, Louisiana
  - Trialspark - Sood, Bowie, Maryland
  - Capital Diabetes and Endocrine Associates, Camp Springs, Maryland
  - Metropolitan Gastroenterology Group PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Woodholme Gastroenterology Associates, P.A., Glen Burnie, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Commonwealth Clinical Studies, PLLC., Brockton, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Synexus Clinical Research US, Inc, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - USMA Clinical Research, LLC, Elizabeth, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Synexus Clinical Research US, Inc., Jamaica, New York
  - Winthrop-University Hospital, Mineola, New York
  - Carolina Digestive Health Associates, PA, Davidson, North Carolina
  - Kinston Medical Specialists, P.A., Kinston, North Carolina
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - Diabetes & Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Synexus Clinical Research US - Cincinnati, Cincinnati, Ohio
  - Synexus Clinical Research US, Inc, Cincinnati, Ohio
  - The MetroHealth System MHS, Cleveland, Ohio
  - Digestive Disease & Surgery Institute, Cleveland, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - CIC America Clinical Inquest Center Ltd., Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Centennial Health-Synexus, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Care Access Research, Warwick, Rhode Island
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinsearch, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - ClinRx Research, LLC, Carrollton, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Biopharma Informatic Inc., Research Center, Houston, Texas
  - Houston Endoscopy and Research Center, Inc., Houston, Texas
  - Rodriguez Clinical Trials, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - Digestive & Liver Disease Center of San Antonio, PLLC, San Antonio, Texas
  - Dwayne O. Williams MD, Sugar Land, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Manassas Clinical Research Centre, Manassas, Virginia
  - VA Medical Center McGuire VAMC, Richmond, Virginia
  - Washington Gastroenterology PLLC, Tacoma, Washington
- Argentina (10):
  - Maffei Centro Medico-Investigacion Clinica Aplicada, C.a.b.a., Buenos Aires
  - Hospital Sirio Libanes, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata SRL, Mar del Plata, Buenos Aires
  - Instituto Privado de Investigaciones Clínicas de Córdoba, Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas de Rosario, Rosario, Santa Fe Province
  - Instituto de Hematologia y Medicina Clinica Dr. Ruben Davoli, Rosario, Santa Fe Province
  - Clinica Mayo - Infectious DiseasesClínica Mayo de Urgencias, San Miguel de Tucumán, Tucumán Province
  - CIPREC, Buenos Aires
  - Centro Universitario de Investigacion en Farmacologia Clinic, Corrientes
  - CIDIM - Centro Integral de Diagnóstico por Imágenes Marchegian, Córdoba
- Austria (4):
  - Ordination, Sankt Stefan, Styria
  - VIVIT Institute, am LKH Feldkirch, Feldkirch, Vorarlberg
  - Privatklinik Wehrle-Diakonissen, Salzburg
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
- Belgium (3):
  - AZ Sint Lucas Brugge, Bruges, Antwerpen
  - Universitair Ziekenhuis Antwerpen, Gastro-Enterologie,, Edegem, Antwerp
  - UZ Brussel, Jette, Brussels Capital
- Brazil (10):
  - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Hospital Universitario Joao de Barros Barreto, Belém, Pará
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto Catarinense de Endocrinologia e Diabetes (ICED), Joinville, Santa Catarina
  - Scentryphar Pesquisa Clinica Ltda, Campinas, São Paulo
  - Instituto de Pesquisa Clinica em Campinas, Campinas, São Paulo
  - CPQuali Pesquisa Clinica Ltda, Santa Cecília, São Paulo
  - Instituto de Estudos E Persquisas Clinicas do Ceará - IEP/CE - Oncology, Fortaleza
  - Instituto de Pesquisa ClÍnica e Medicina AvanCada Ltda, São Paulo
- Canada (14):
  - University of Calgary, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - CISSS de la Monteregie-Centre, Greenfield Park, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CHUM, Montreal, Quebec
  - Central Alberta Research Centre, Red Deer
- Colombia (11):
  - Centro Cardiovascular Colombiano Clínica Santa María, Medellín, Antioquia
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Centro Cardiovascular y de Diabetes, Barranquilla, Atlántico
  - Fundacion Bios, Barranquilla, Atlántico
  - Medplus Mp, Bogotá, Bogota D.C.
  - Endocare Ltda., Bogotá, Bogota D.C.
  - Asociación Colombiana de Diabetes, Bogotá, Cundinamarca
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Fundacion Centro de Investigaciones Clinicas CARDIOMET, Pereira, Risaralda Department
  - IPS Centro Medico Julian Coronel S.A, Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A., Cali, Valle del Cauca Department
- Denmark (3):
  - Gastroenheden, Hvidovre hospital, Hvidovre, Copenhagen
  - Endocrinology, Aalborg University Hospital, Aalborg
  - Center for Clinical Metabolic Research, Hellerup
- Germany (7):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-SWÃƒÂ¼rttemberg
  - Studienzentrum Schwittay, Böhlen, Saxony
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Clinical Research Unit, Giessen
  - Clinical Research Hamburg, Hamburg
  - Israelitisches Krankenhaus, Hamburg
  - KRH Klinikum Siloah, Hanover
- Hungary (10):
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger, Heves County
  - BKS Research Kft Synexus AS, Hatvan, Heves County
  - Hetenyi Geza Hospital, Szolnok, Jász-Nagykun-Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg, Zala County
  - Synexus Budapest DRS, Budapest
  - Strázsahegy Gyógyszertár Medicina, Budapest
  - SYNEXUS Magyarorszag Kft Debrecen A.S., Debrecen
  - Synexus Magyarország kft. Gyula DRS, Gyula
  - Szegedi Tudomanyegyetem, Szeged
  - Synexus Magyarorszag Kft, Zalaegerszeg
- Latvia (4):
  - Polana-D, Daugavpils
  - Kraslava Hospital, Krāslava
  - Pauls Stradins Clinical University Hospital, Endokrinologijas nodala, Riga
  - Digestive Diseases Centre GASTRO, Riga
- Mexico (12):
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Consultorio Medico, Guadalajara, Jalisco
  - Unidad de Investigación Clínica en Medicina S.C., Guadalajara, Jalisco
  - Medical and Nutritional Trials, Cuauhtémoc, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevencion de E - Endocrinology, Mexico City, Mexico City
  - Centro de Atención e Investigación en Factores de Riesgo Car, Mexico City, Mexico City
  - Clinicos Asociados BOCM SC, Portales, Mexico City
  - Centro de Desarrollo Biomedico S.C.P., Mérida, Yucatán
  - Centro de Investigacion Cardiometabolica de Aguascalientes SA de CV, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Dioderm Instituto de Investigacion, Durango
  - Sociedad de Metabolismo y Corazon, S.C., Veracruz
- Russia (11):
  - Saint-Petersburg City Pokrovskaya Hospital, St-Petersburg, Leningradskaya Oblast'
  - Scientific Institute of Clinical and Experimental Lymphology, Novosibirsk, Novosibirsk Oblast
  - GUZ Saratov City Clinical Hospital 9, Saratov, Saratov Oblast
  - Nizhegorodsky Regional Clinical Hospital named after N. A. Semashko, Nizhny Novgorod, Volga
  - Kazan State Medical University, Kazan'
  - FSBI National medical endocrinology research centre, Moscow
  - Moscow Regional Research Clinical Institute named by MF Vladimirski, Moscow
  - Rostov on Don, Rostov-on-Don
  - Rostov State Medical University, Rostov-on-Don
  - North-Western State Medical University named after I. I. Mechnikov, Saint Petersburg
  - Saratov City Clinical Hospital 12, Saratov
- South Africa (6):
  - FARMOVS, Bloemfontein, Free State
  - Wits Clinical Research, Johannesburg, Gauteng
  - Synexus Stanza Clinical Research Centre, Pretoria, Gauteng
  - Watermeyer Clinical Research Site, Silverton, Gauteng
  - Synexus Helderberg Clinical Research Centre, Cape Town, Western Cape
  - TREAD Research, Cape Town
- United Kingdom (21):
  - MAC Clinical Research Manchester, Manchester, Greater Manchester
  - Synexus Lancashire Dedicated Research Centre, Chorley, Lancashire
  - Royal Oldham Hospital, Oldham, Lancashire
  - MAC Research, Exchange House, Cannock, Staffordshire
  - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands
  - MAC Clinical Research, Monarch House, Leeds, West Yorkshire
  - MAC Research, Barnsley
  - MAC Clinical Research, Blackpool
  - Synexus Wales Clinical Research Centre, Cardiff
  - Mid Essex Hospital Services NHS Trust Broomfield Hospital, Chelmsford
  - Western General Hospital, Edinburgh
  - Synexus Merseyside Dedicated Research Centre, Liverpool
  - MAC Clinical Research, Liverpool
  - Wingate Institute of Neurogastroenterology and Barts Health Trust and the Royal London Hospital, London
  - MAC Clinical Research, GAC House, Manchester
  - Synexus Manchester Clinical Research Centre, Manchester
  - Royal Victoria Infirmary: Clinical Research Facility, Newcastle upon Tyne
  - Biomedical Research Centre, Nottingham
  - Synexus Hexham Dedicated Research Centre, Stockton-on-Tees
  - Synexus North Tees Clinical Research Centre, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Relamorelin 10 μg
Started | 155 | 156
Safety Population (The Safety Population included all participants who received ≥1 administration of double-blind study treatment.) | 152 | 155
Completed | 137 | 139
Not Completed | 18 | 17
Not completed — Adverse Event | 4 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Deviation | 3 | 4
Not completed — Reason Not Specified | 1 | 2
Not completed — Missing Completion Status | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Relamorelin 10 μg: Following a 2-week placebo run-in, participants received relamorelin 10 μg injected subcutaneously twice daily for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Relamorelin 10 μg | Total
Number analyzed (Participants) | 155 | 156 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.13) | 55.8 (12.07) | 55.0 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 114 | 226
  Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 51 | 105
  Not Hispanic or Latino | 101 | 105 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 11
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 17 | 42
  White | 123 | 127 | 250
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Diabetic Gastroparesis Symptom Severity Score (DGSSS)
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the Diabetic Gastroparesis Symptom Severity Diary (DGSSD), recorded in an electronic diary (e-diary). The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0= no or not at all uncomfortable to 10= worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period.
Time Frame: Baseline (Day-14 to Day-1) to Week 12
Population: Modified Intent-to-treat (mITT) Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
score on a scale
  Baseline | 23.4 (5.40) | 24.9 (6.15)
  Change from Baseline to Week 12 | -9.3 (10.21) | -10.2 (9.24)

2. Primary Outcome: Percentage of Participants Meeting the Vomiting Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. A Vomiting Responder was defined as a participant with zero weekly vomiting episodes during each of the last 6 weeks of the 12-week Treatment Period.
Time Frame: Week 6 to Week 12
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
percentage of participants | 19.1 | 18.7

3. Secondary Outcome: Percentage of Participants Meeting the Nausea Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Nausea Responder was defined as a participant with improvement (decrease) of at least 2-points in the weekly symptom scores for nausea at each of the last 6 weeks of the 12-week Treatment Period. Nausea was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0= no nausea to 10= worst possible nausea.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
percentage of participants | 32.9 | 38.1

4. Secondary Outcome: Percentage of Participants Meeting the Abdominal Pain Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: An Abdominal Pain Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for abdominal pain at each of the last 6 weeks of the 12-week Treatment Period. Abdominal pain was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0= no abdominal pain to 10= the worst possible abdominal pain and was recorded in an e-diary.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
percentage of participants | 27.0 | 36.1

5. Secondary Outcome: Percentage of Participants Meeting the Bloating Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Bloating Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for bloating at each of the last 6 weeks of the 12-week Treatment Period. Bloating was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0= no bloating and 10= the worst possible bloating and was recorded in the e-diary.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
percentage of participants | 27.0 | 31.6

6. Secondary Outcome: Percentage of Participants Meeting the Postprandial Fullness Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Postprandial Fullness Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for Postprandial Fullness at each of the last 6 weeks of the 12-week Treatment Period. Postprandial Fullness was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0= no feeling of fullness until finishing a meal (best) to 10= feeling full after only a few bites (worst).
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
percentage of participants | 23.7 | 27.7

7. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is an AE that begins or worsens after receiving study drug.
Time Frame: Up to approximately 16 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
Participants | 75 | 86

8. Secondary Outcome: Number of Participants With Potential Clinically Significant (PCS) Clinical Laboratory Results
Description: Clinical Laboratory tests included Hematology, Chemistry and Urinalysis tests. The investigator determined if the results were clinically significant. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment. Number analyzed is the number of participants with non-PCS baseline values and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
Participants
  Eosinophils Absolute Cell Count [10^9/liter (L)]: >3×Upper Limit of Normal Value (ULN): number analyzed (Participants) | 144 | 152
  Eosinophils Absolute Cell Count [10^9/liter (L)]: >3×Upper Limit of Normal Value (ULN) | 0 | 1
  Hematocrit (RATIO): >1.1×ULN: number analyzed (Participants) | 137 | 149
  Hematocrit (RATIO): >1.1×ULN | 1 | 0
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN): number analyzed (Participants) | 137 | 149
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN) | 4 | 4
  Hemoglobin [grams (g)/L]: <0.9×LLN: number analyzed (Participants) | 134 | 148
  Hemoglobin [grams (g)/L]: <0.9×LLN | 2 | 5
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 141 | 148
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN | 1 | 3
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN: number analyzed (Participants) | 142 | 151
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN | 1 | 1
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 142 | 148
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN | 0 | 1
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 142 | 148
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN | 2 | 2
  Red Blood Cell Count (10^12/L): <0.9×LLN: number analyzed (Participants) | 139 | 150
  Red Blood Cell Count (10^12/L): <0.9×LLN | 1 | 1
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN: number analyzed (Participants) | 146 | 151
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN | 1 | 0
  Albumin (g/L): <0.9×LLN: number analyzed (Participants) | 145 | 152
  Albumin (g/L): <0.9×LLN | 0 | 1
  Alkaline Phosphatase (U/L): >=3×ULN: number analyzed (Participants) | 146 | 152
  Alkaline Phosphatase (U/L): >=3×ULN | 1 | 0
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN: number analyzed (Participants) | 146 | 152
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN | 1 | 2
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN: number analyzed (Participants) | 142 | 145
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN | 0 | 1
  Bicarbonate (HCO3) (mmol/L): <0.9×LLN: number analyzed (Participants) | 142 | 145
  Bicarbonate (HCO3) (mmol/L): <0.9×LLN | 1 | 0
  Blood Urea Nitrogen (mmol/L): >1.2×ULN: number analyzed (Participants) | 130 | 133
  Blood Urea Nitrogen (mmol/L): >1.2×ULN | 15 | 3
  Chloride (mmol/L): <0.9×LLN: number analyzed (Participants) | 146 | 152
  Chloride (mmol/L): <0.9×LLN | 2 | 0
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN: number analyzed (Participants) | 139 | 148
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN | 2 | 1
  Creatinine [micromoles(μmol)/L]: >1.3×ULN: number analyzed (Participants) | 132 | 142
  Creatinine [micromoles(μmol)/L]: >1.3×ULN | 8 | 7
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN: number analyzed (Participants) | 124 | 132
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN | 11 | 21
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN: number analyzed (Participants) | 124 | 132
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN | 6 | 5
  Glycohemoglobin A1C: Increase of >=0.5%: number analyzed (Participants) | 146 | 151
  Glycohemoglobin A1C: Increase of >=0.5% | 80 | 111
  Glycohemoglobin A1C: Increase of >=1%: number analyzed (Participants) | 146 | 151
  Glycohemoglobin A1C: Increase of >=1% | 80 | 111
  Phosphorus (mmol/L): >1.1×ULN: number analyzed (Participants) | 142 | 147
  Phosphorus (mmol/L): >1.1×ULN | 5 | 5
  Phosphorus (mmol/L): <0.9×LLN: number analyzed (Participants) | 142 | 147
  Phosphorus (mmol/L): <0.9×LLN | 1 | 1
  Potassium (mmol/L): <0.9×LLN: number analyzed (Participants) | 146 | 152
  Potassium (mmol/L): <0.9×LLN | 1 | 0
  Sodium (mmol/L): <0.9×LLN: number analyzed (Participants) | 146 | 152
  Sodium (mmol/L): <0.9×LLN | 1 | 0
  Triglycerides, Fasting (mmol/L): >=3×ULN: number analyzed (Participants) | 137 | 144
  Triglycerides, Fasting (mmol/L): >=3×ULN | 3 | 5
  Uric Acid (Urate) (μmol/L): >1.1×ULN: number analyzed (Participants) | 125 | 121
  Uric Acid (Urate) (μmol/L): >1.1×ULN | 18 | 13
  Uric Acid (Urate) (μmol/L): <0.9×LLN: number analyzed (Participants) | 125 | 121
  Uric Acid (Urate) (μmol/L): <0.9×LLN | 3 | 0

9. Secondary Outcome: Number of Participants With Clinically Meaningful Trends for Vital Signs
Description: Vital Signs included assessments of heart rate, respiratory rate, systolic and diastolic blood pressure, and body temperature. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results
Description: A standard 12-lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 152 | 155
Participants | 1 | 2

11. Secondary Outcome: Number of Participants With a ≥1% Increase in Glycosylated Hemoglobin A1c (HBA1c)
Time Frame: Baseline (Day 1) up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment. Overall number analyzed is the number of participants with non-PCS baseline values and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 146 | 151
Participants | 80 | 111

12. Secondary Outcome: Number of Participants With Anti-relamorelin Antibody Testing Results by Visit
Description: A blood sample was collected that was sent to a laboratory for an anti-relamorelin antibody screening test. A positive screening test was confirmed by an immunodepletion assay. The number of participants in each of the following categories are reported: Negative Screening Test, Positive Screening Test, Negative Confirmatory Test, and Positive Confirmatory Test at each time point.
Time Frame: Baseline (Day 1), Day 14, Day 28, Day 84, and End of Treatment (Up to Day 84)
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment (N=155 in the Relamorelin 10 μg arm). Anti-relamorelin antibody testing was only done for those participants who received treatment with relamorelin. Number analyzed is the number of participants with data available at the given timepoint. Due to a laboratory issue not all positive screening tests were confirmed.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin 10 μg
Number analyzed (Participants) | 155
Participants
  Screening Test (Baseline): number analyzed (Participants) | 145
  Screening Test (Baseline): Negative | 127
  Screening Test (Baseline): Positive | 18
  Confirmatory Test (Baseline): number analyzed (Participants) | 12
  Confirmatory Test (Baseline): Negative | 12
  Confirmatory Test (Baseline): Positive | 0
  Screening Test (Day 14): number analyzed (Participants) | 133
  Screening Test (Day 14): Negative | 115
  Screening Test (Day 14): Positive | 18
  Confirmatory Test (Day 14): number analyzed (Participants) | 13
  Confirmatory Test (Day 14): Negative | 13
  Confirmatory Test (Day 14): Positive | 0
  Screening Test (Day 28): number analyzed (Participants) | 121
  Screening Test (Day 28): Negative | 104
  Screening Test (Day 28): Positive | 17
  Confirmatory Test (Day 28): number analyzed (Participants) | 12
  Confirmatory Test (Day 28): Negative | 12
  Confirmatory Test (Day 28): Positive | 0
  Screening Test (Day 84): number analyzed (Participants) | 104
  Screening Test (Day 84): Negative | 87
  Screening Test (Day 84): Positive | 17
  Confirmatory Test (Day 84): number analyzed (Participants) | 12
  Confirmatory Test (Day 84): Negative | 11
  Confirmatory Test (Day 84): Positive | 1
  Screening Test (End of Treatment): number analyzed (Participants) | 7
  Screening Test (End of Treatment): Negative | 6
  Screening Test (End of Treatment): Positive | 1
  Confirmatory Test (End of Treatment): number analyzed (Participants) | 1
  Confirmatory Test (End of Treatment): Negative | 1
  Confirmatory Test (End of Treatment): Positive | 0
  Screening Test (Unscheduled): number analyzed (Participants) | 6
  Screening Test (Unscheduled): Negative | 6
  Screening Test (Unscheduled): Positive | 0
  Positive Confirmatory Test (Unscheduled): number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 16 weeks
Description: All-Cause Mortality is reported for all randomized participants. The Safety Population, all participants who received ≥1 administration of double-blind study treatment, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Relamorelin 10 μg
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/156
Serious Adverse Events (participants affected / at risk) | 6/152 | 8/155
Other Adverse Events (participants affected / at risk) | 14/152 | 13/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=152) | Relamorelin 10 μg (N=155)
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/109 | 1/113 — Number at risk is based on the female population.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=152) | Relamorelin 10 μg (N=155)
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Urinary tract infection (Infections and infestations) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03426345/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03426345/SAP_001.pdf